CLINICAL TRIAL: NCT07284615
Title: Lateral Femoral Cutaneous Nerve (LFCN) Block or Wound Infiltration (WI) Combined With Pericapsular Nerve Group (PENG) Block for Analgesia in Elective Anterior Approach Total Hip Arthroplasty: A Randomized Controlled Trial
Brief Title: Pericapsular Nerve Group (PENG) Block Combined With Lateral Femoral Cutaneous Nerve (LFCN) Block or Wound Infiltration for Postoperative Analgesia in Anterior Approach Total Hip Arthroplasty: A Randomized Controlled Trial
Acronym: Peng_lfcn/WI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale Edoardo Bassini (Other)
Responsible Party: Principal Investigator, Matteo Coccolo, Medical Doctor, Principal Investigator, Ospedale Edoardo Bassini
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5967
Record Dates: First submitted 2025-11-19; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Arthropathy of Hip; Hip Arthropathy; Locoregional Anesthesia; Complication of Anesthesia; Regional Anesthesia Morbidity; Hospital Stay, Length of Stay in Hospital From Time of Surgery Till Discharge; Opioid Consumption
Keywords: Postoperative muscle weakness; ERAS; Regional Block

STUDY DESIGN:
Intervention Model Description: A double-blind, randomized, controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The anesthetist in the operating room will be the only one who knows what treatment has been administered
  Participant: the patient will not know the type of block he will be subjected to, because of he will already be subjected to neuraxial anesthesia.
  Outcomes Assessor: a clinician external to the practice will evaluate the degree of residual paralysis after anesthesia and pain control Investigator: the statistician will not know which anesthetic technique was administered to which group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG - LFCN Block (Experimental): group in which PENG and LFCN Block was performed. After performing neuraxial anesthesia, the PENG associated with LFCN block will be performed. Under ultrasound guidance, 20ml and 10ml of Ropivacaine 0.5% will be administered respectively
  Interventions: Procedure: PENG plus LFCN block
- PENG-WI (Active Comparator): the group in which PENG and WI (wound infiltration) are performed, after neuraxial anesthesia, a PENG block will be administered under ultrasound guidance using 20 mL of 0.5% ropivacaine. At the end of the surgery, a wound infiltration will be performed with 10 mL of 0.5% ropivacaine.
  Interventions: Procedure: PENG plus WI

INTERVENTIONS:
Procedure: PENG plus LFCN block — The experimental arm will be subjected to a combination of peripheral blocks: the interfascial block of the PENG and the perinervous block of the LFCN The PENG block involves deposition of local anesthetic in the fascial plane between the psoas muscle and the superior pubic ramus. The LFCN block consists of applying local anesthetic near the nerve. The LFCN lies in the subcutaneous plane deep to the fascia lata below the anterior superior ischiatic spine.
  Other Names: Pericapsular nerve group block and lateral femoral cutaneous nerve block, PENG and lateral femoral cutaneous nerve block
  Arms: PENG - LFCN Block
Procedure: PENG plus WI — The control arm will receive a combination of pericapsular nerve group (PENG) block and wound infiltration (WI). The PENG block involves the deposition of local anesthetic in the fascial plane between the psoas tendon and the superior pubic ramus, under ultrasound guidance. The wound infiltration consists of the administration of local anesthetic into the subcutaneous tissue along the surgical incision
  Other Names: Pericapsular nerve group block and wound infiltration, PENG and WI
  Arms: PENG-WI

SUMMARY:
This prospective, randomized controlled trial aims to compare two multimodal regional anesthesia strategies for postoperative analgesia in elective total hip arthroplasty (THA) performed via anterior approach. Patients will be randomized to receive either a Pericapsular Nerve Group (PENG) block combined with a Lateral Femoral Cutaneous Nerve (LFCN) block, or a PENG block combined with wound infiltration (WI).

The primary outcome is postoperative pain intensity at rest, measured by Numerical Rating Scale (NRS) at 6 hours after surgery. Secondary outcomes include dynamic pain scores at 6, 24, and 48 hours, total opioid consumption, time to first rescue analgesia, quadriceps strength, hip flexion angle, length of stay, and adverse events.

All procedures are routinely used in clinical practice and carry minimal additional risk. Safety will be continuously monitored by the Principal Investigator and the study team according to an internal Safety Monitoring Plan.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Elective total hip arthroplasty
* Spinal (subarachnoid) anesthesia
* Written informed consent provided by the patient or by the legal guardian, if appointed

Exclusion Criteria:

* INR > 1.5
* aPTT > 1.5
* Platelet count < 75,000/mm³
* Signs suggestive of infection at the puncture site
* Absence of informed consent to the procedure
* Documented or suspected allergy to local anesthetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Pain at rest control at 6h | six hours after performing the regional anesthesia technique
  pain assessment with Numeric Rating Scale (NRS): a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"

SECONDARY OUTCOMES:
Pain at rest control at 24h | 24 hours after performing the regional anesthesia technique
  pain assessment with Numeric Rating Scale (NRS): a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"
Pain at rest control at 48h | 48 hours after performing the regional anesthesia technique
  pain assessment with Numeric Rating Scale (NRS): a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"
Pain on movement control at 6h | six hours after performing the regional anesthesia technique
  pain assessment with Numeric Rating Scale (NRS): a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"
Pain on movement control at 24h | 24 hours after performing the regional anesthesia technique
  pain assessment with Numeric Rating Scale (NRS): a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"
Pain on movement control at 48h | 48 hours after performing the regional anesthesia technique
  pain assessment with Numeric Rating Scale (NRS): a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"
MRC at 6h | six hours after performing the regional anesthesia technique
  evaluation of the degree of weakness or residual paresis of the quadriceps femoris muscle on the operative side using 'the Oxford Scale' (aka Medical Research Council Manual Muscle Testing scale or MRC scale) The MRC scale is a 0-5 scale, with zero meaning "no contraction " and five meaning "Full range of motion against gravity with full resistance".
MRC at 24h | 24 hours after performing the regional anesthesia technique
  evaluation of the degree of weakness or residual paresis of the quadriceps femoris muscle on the operative side using 'the Oxford Scale' (aka Medical Research Council Manual Muscle Testing scale or MRC scale) The MRC scale is a 0-5 scale, with zero meaning "no contraction " and five meaning "Full range of motion against gravity with full resistance".
MRC at 48h | 48 hours after performing the regional anesthesia technique
  evaluation of the degree of weakness or residual paresis of the quadriceps femoris muscle on the operative side using 'the Oxford Scale' (aka Medical Research Council Manual Muscle Testing scale or MRC scale) The MRC scale is a 0-5 scale, with zero meaning "no contraction " and five meaning "Full range of motion against gravity with full resistance".
time to first PRN opioid request | Time Frame: From date of surgery until up to 48 hours after
  Description: time to first PRN (pro re nata) opioid request expressed in minutes
MME of PRN opioid total doses | From date of surgery until up to 48 hours after
  Description: Morphine Milligram Equivalents (MME) of "pro re nata" (PRN) opioid total doses we will study the effect of Regional anesthesia on opioid-sparing with the same pre-established pain relief protocol
Complication | From date of surgery until up to 48 hours after
  any complications recorded in the first 48 hours including but not limited to: postoperative nausea and vomiting (PONV), vascular puncture, paresthesia and LA toxicity
the degree of hip flexion at 6h | six hours after performing the regional anesthesia technique
  Hip flexion degree of the operative side is measured using Digital Angle Gauge in supine position
the degree of hip flexion at 24h | 24 hours after performing the regional anesthesia technique
  Hip flexion degree of the operative side is measured using Digital Angle Gauge in supine position
the degree of hip flexion at 48h | 48 hours after performing the regional anesthesia technique
  Hip flexion degree of the operative side is measured using Digital Angle Gauge in supine position
Length of Hospital Stay (LOS) | From date of surgery until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 10 months
  Length of hospital stay will be recorded as the number of postoperative midnights spent in the Orthopedic Ward, calculated from the day of surgery (postoperative day 0) until the date of discharge or death (exitus).

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Edoardo Bassini, Cinisello Balsamo, Milano, Italy

IPD SHARING:
Plan to Share IPD: No